CLINICAL TRIAL: NCT04242108
Title: Diagnostic Performance of Deep Convolutional Neural Networks for Angle Closure Glaucoma: an International Multicenter Study
Brief Title: Diagnostic Performance of Deep Learning for Angle Closure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2018KYPJ074
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Angle Closure Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Angle closure group
  Interventions: Diagnostic Test: Deep learning algorithm based on AS-OCT scans
- Open angle group
  Interventions: Diagnostic Test: Deep learning algorithm based on AS-OCT scans
- Peripheral synechia (PAS) group
  Interventions: Diagnostic Test: Deep learning algorithm based on AS-OCT scans
- Non-peripheral synechia (PAS) group
  Interventions: Diagnostic Test: Deep learning algorithm based on AS-OCT scans

INTERVENTIONS:
Diagnostic Test: Deep learning algorithm based on AS-OCT scans — The OCT scans of study subjects would be imported into the algorithm. Automated classfication of angle width and detection of synechia would be performed by the algorithm. The diagnostic performance of the algorithm would be compared with gonioscopy records.

SUMMARY:
Primary angle closure diseases (PACD) are commonly seen in Asia. In clinical practice, gonioscopy is the gold standard for angle width classification in PACD patietns. However, gonioscopy is a contact examination and needs a long learning curve. Anterior segment optical coherence tomography (AS-OCT) is a non-contact test which can obtain three dimensional images of the anterior segment within seconds. Therefore, the investigators designed the study to verify if AS-OCT based deep learning algorithm is able to detect the PACD subjects diagnosed by gonioscopy.

ELIGIBILITY:
The inclusion criteria in the study were as follows: (1) All participants must be ≥ 18 years old; (2) Study subjects had a previous diagnosis of the ACA status (narrow or open, PAS or non-PAS) based on gonioscopy, SS-OCT scans and medical history records. Exclusion criteria of the data include: (1) poor compliance in receiving gonioscopy examination; (2) unclear AS-OCT scans due to blinking or out of focus; (3) recent use of miotics within a month; 4) secondary angle closure sue to subluxation or dislocation, uveitis, neovascular glaucoma, et al.; 5) history of ocular surgery or laser iridotomy; 6) patients who previously had an episode of primary angle closure (which was obtained on history by asking the patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The training and primary validation datasets were collected from the databases of electronic medical and research records at Zhongshan Ophthalmic Center from September 1, 2016, to September 1, 2019. The external test dataset was obtained from the Singapore Eye Research Institute (SERI), Singapore during June 2008 to November 2019, and the Chulalongkorn University and King Chulalongkorn Memorial Hospital (KCMH, Bangkok, Thailand) from October, 2019 to April, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Area under receiver operating curve (AUC) | Immediately after obtaining the AS-OCT images
  AUC value of the deep learning algorithm in angle width classfication and synechia detection

SECONDARY OUTCOMES:
Sensitivity and specificity | Immediately after obtaining the AS-OCT images
  Sensitivity and specificity of the automated algorithm in angle width classfication and synechia detection

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The imaging data of study subjects would be available to other researchers upon reasonable request. Part of the data would be open as public datasets after the related article is published.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Part of the data would be open as public datasets after the related article is published.